CLINICAL TRIAL: NCT06509490
Title: A Single-center, Open, Single-arm Clinical Study of the Safety and Efficacy of KD-025 CAR-T Therapy in Advanced NKG2DL+ Solid Tumors
Brief Title: NKG2D CAR-T(KD-025) in the Treatment of Advanced NKG2DL+ Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NING_LI, Associate President, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD-025-XJM
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Safety Issues

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KD025 (Experimental): This group of patients received KD025 cell injection.
  Interventions: Drug: KD-025 cell injection

INTERVENTIONS:
Drug: KD-025 cell injection — This is an open-label, dose escalation/expansion study to assess the safety, tolerability, and efficacy of KD-025 cell infusion in patients with advanced NKG2DL+ solid tumor. In this study,the enrollment of the patients must meet the inclusion and exclusion criteria . All subjects will be undergo screening, pre-treatment (cell product preparation;lymphodepleting chemotherapy), treatment and follow up

SUMMARY:
This is a Phase 1, single-arm, single-center, open-label study to evaluate the safety and effectiveness of NKG2D-based CAR-T cells infusion in the treatment of advanced NKG2DL+ solid tumors.

DETAILED DESCRIPTION:
This is an open-label, dose escalation/expansion study to assess the safety, tolerability, and efficacy of KD-025 cell infusion in patients with advanced NKG2DL+ solid tumor. In this study,the enrollment of the patients must meet the inclusion and exclusion criteria . All subjects will be undergo screening, pre-treatment (cell product preparation;lymphodepleting chemotherapy), treatment and follow up

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as advanced solid tumors histopathologically or cytologically, such as ovarian, cholangiocarcinoma, and colorectal cancer.
2. Patients fail standard treatment , or cannot tolerate standard treatment, or there is no standard treatment, the standard treatment recommendations refer to the latest version of the guidelines of the national comprehensive cancer network (NCCN) or the guidelines of the Chinese society of Clinical Oncology (CSCO);
3. Age 18-70 years;
4. ECOG score 0-1;
5. Expected survival ≥ 3 months;
6. Patients must meet coagulation parameters and have adequate peripheral venous access for apheresis, and must also have enough PBMC to manufacture CAR T cells;
7. NKG2DL (according to the positive comprehensive score of 0-12 points, positive SCORE of NKG2DL ≥2) positive confirmed byImmunohistochemistry. Biopsy tissue must be no more than 1 year, if not, must obtain new tissue material from a recent surgical or diagnostic biopsy;
8. Eligible organ and bone marrow functions defined as follows:1) Absolute neutrophil count ≥1.5×10^9/L, lymphocyte count ≥0.5×10^9/ L, platelet count ≥90×10^9/L, hemoglobin ≥90g/L (no blood transfusion or Erythropoietin within 7 days); 2) Total bilirubin ≤2ULN; Serum alanine amino transferase (ALT) or aspartate aminotransferase (AST)≤2.5ULN (≤2.5 times with liver metastasis); 3) Creatinine ≤1.5ULN or eGFR≥ 60mL /min/1.73m^2 [eGFR=186×(age)-0.203×SCr-1.154(mg/dl), eGFR timing in women was 0.742]; 4) International normalized ratio (INR) or prothrombin time (PT) ≤1.5ULN; 5) Lung function: ≤ grade 1 dyspnea (according to NCI-CTCAE V5.0), SaO2≥91%; 6) Cardiac function: Cardiac ejection fraction (LVEF) detected by echocardiography or MUGA ≥50% 1 month before enrollment.
9. Patients must have measurable lesions as defined by RECIST 1.1;
10. Patients fully understand the test and voluntarily sign the informed consent;
11. Patient agree to use approved contraceptive methods (e.g., birth control pills, barrier devices, iuds, contraindicated drugs) during the study and for at least 12 months after last cell infusion, until no CAR-T cells were detected by two consecutive PCR tests.

Exclusion Criteria:

1. Patients had received any gene therapy (including CAR-T cell therapy) or any T cell therapy, Active bacteria or viral or fungal infection and not controlled after anti-infective treatment (positive blood test 72 hours before infusion), Syphilis, Human immunodeficiency virus (HIV), Active hepatitis B (HBV DNA≥500IU/ml) or hepatitis c (anti-HCV positive and HCV RNA higher than the detection limit of analysis method);
2. Patients have an autoimmune disease or organ transplant, require chronic systemic steroid therapy or any other form of immunosuppressive drugs;
3. A history of serious heart or lung disease, including uncontrolled hypertension medication, and any condition that occurred within the past 6 months: congestive heart failure (New York Heart Association functional classification ≥3), cardiac angioplasty and stents, myocardial infarction, unstable angina, or other clinically severe heart disease;
4. Detected clinically relevant central nervous system (CNS) metastases and/or pathologies, such as seizures, cerebral ischemia/bleeding, dementia, cerebellar diseases or autoimmune diseases affecting the CNS;
5. The Patients' history or existing evidence of any condition such as neuroticism, psychosis, immunology, metabolism, and infectious disease, in any treatment, or laboratory abnormalities may confuse the outcome of the study, interfere with the Patients' participation during the study, or not participate in the Patients' best interests with investigator treatment;
6. The Patients have a history of hematologic malignancy or concurrent history of other malignant primary solid tumors, except for: 1) Patients with cervical or breast cancer in situ who have no evidence of disease for more than 3 years after radical treatment; 2) Patients who have successfully received definite resection of tumor in situ and have no evidence of disease for ≥5 years;
7. Received chemotherapy, radiation, small molecule, biologic cancer therapy, immunotherapy, or other experimental drugs within 4 weeks prior to study initiation,
8. Pregnant or lactating women;
9. The investigator considers the Patients have or with current historical evidence of any condition, therapy, or laboratory anomaly that may confound the results of the study, interfere with the Patients' participation in the fulltime study and the requirements of the cooperative trial, not controlled medical, psychological, family, social, or geographic conditions, or not participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-07-17 (Estimated); Primary Completion 2024-07-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
treatment-emergent adverse events(TEAEs) | 3 months after single infusion
  An adverse event is any undesirable experience associated with the use of a medical product in a patient
Dose-limiting toxicity (DLT) rate | 3 months after single infusion
  A drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose.
CAR positive T cells in patients | 6 months after single infusion
  The time of CAR-T cell reach the peak and turn back to baseline

SECONDARY OUTCOMES:
Objective response rate(ORR) | 1month,2month,3month,6month,1 year after cell infusion]
  objective tumor response rate will be calculated for patients with measurable disease per RECIST 1.1 only
Progression free survival(PFS) | 1month,2month,3month,6month,1 year after cell infusion]
  the time from the date of first infusion of the KD-025 to the first documented disease progression (according to RECIST 1.1) or death (due to any cause), whichever occurs first
Overall survival #OS# | 1month,2month,3month,6month,1 year after cell infusion
  the time from the date of first infusion of KD-025 to death of the subject
Complete remission (CR) | 1month,2month,3month,6month,1 year after cell infusion
  the time from the date of first infusion of KD-025 to death of the subject

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Principal Investigator — NCCICAMS
Locations (1):
- Cancer hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No